CLINICAL TRIAL: NCT02958800
Title: Developing a Single Patient Open-label Trial Tapering Algorithm for Antipsychotics in Long-Term Care - A Pilot Study
Brief Title: Deprescribing Antipsychotics in Long-Term Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: College of Family Physicians of Canada (Other); MediSystem Pharmacy (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CFPC-86796210
Record Dates: First submitted 2016-11-02; First posted 2016-11-08 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Dementia; Behavior
Keywords: Deprescribing; Single patient open label trial; Long-term care
MeSH Terms: conditions — Dementia; Behavior | interventions — Methods; Risperidone; Quetiapine Fumarate; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): The intervention consists of assigning each participant to their own single patient open label trial consisting of a 1:1 randomized sequence of two pre-determined dose reductions of atypical antipsychotics for each participant in order to determine any behavioural issues that arise from atypical antipsychotic dose alteration.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — The intervention will be 12-weeks in duration consisting of four blocks resulting from a 1:1 randomization of two different three-week treatment courses of a patient's existing antipsychotic medication. For example, the intervention "ABAB" means that a participant would undergo three weeks of treatment A, followed by three weeks of treatment B, followed by three weeks of treatment A, and lastly three weeks of treatment B.
  Treatment A block is defined as a mutually agreed upon dose of a participant's antipsychotic medication that is different (i.e. lower) than their enrolment dose.
  Treatment B block is defined as a mutually agreed upon dose of a participant's antipsychotic medication that is different (i.e. lower) than their enrolment dose and the dose in Treatment A.
  Other Names: Antipsychotic Atypical; Risperidone; Quetiapine; Olanzapine

SUMMARY:
Aggressive behaviours in long-term care (LTC) is a difficult health care issue to manage. One method that has been over-used is the prescription of antipsychotics for the behaviours and psychological symptoms of dementia (BPSD). This high prevalence of use is a recognized health care problem in Ontario and around the world; increased antipsychotics use is associated with increased falls and mortality. Existing strategies are educational in nature and are not systematic; the goal of this study is to develop a systematic algorithm to help LTC physicians deprescribe and taper antipsychotics safely and effectively.

The objectives of the study is to: 1) Develop a discontinuation algorithm for antipsychotics based on single patient open-label (SPOT) trial methodology (e.g. a variation of N-of-1 trials) with standardized outcome measures for LTC physicians; 2) To pilot a clinical pharmacist-led recruitment strategy; 3) To provide preliminary evidence to demonstrate that this algorithm could lead to deprescribing of anti-psychotic medications in LTC.

DETAILED DESCRIPTION:
This pilot study will consist of enrolling long-term care (LTC) patients to a 12-week, single-patient, open-label, randomized multiple crossover trial consisting of 2 different treatment blocks (Block A, Block B) of 3 weeks duration each.

This study is targeting LTC residents in two Hamilton LTC facilities associated with MediSystem pharmacy. Once potential participants have been identified by the clinical pharmacist working at these two facilities, a invitation letter with a consent letter will be sent to the LTC resident's power of attorney for health care (POA-HC) describing the study and inviting them to complete the mail back the consent form. POA-HCs will be provided with contact information of the research assistant associated with the study in order to have any of their questions answered.

Once consent is received, the LTC patient will be assigned a randomized 1:1 treatment sequence of Block A (denoted by "A") and Block B (denoted by "B"). For example, Patient1 may be assigned the treatment sequence AABB, while Patient2 may be assigned the treatment sequence BAAB, and so on. The patient will then take a pre-determined dose, DOSE-A, of the antipsychotic that has been agreed upon between the physician and the POA-HC at time of enrolment during Block A. This pre-determined dose will be less than the current dose the LTC patient is taking at the time of enrolment. Similarly, the LTC patient will take DOSE-B, a second pre-determined dose of the antipsychotic that is different than the starting dose or DOSE-A, will be taken during Block B.

At the end of the 12-week study, LTC physicians will be given a report which describes and summarizes the outcome measures for each participating LTC patient. This report will be reviewed together with the POA-HC in order to make a clinical decision together on whether to continue using the antipsychotic medication, or whether a decreased or discontinued dose is more appropriate. After this decision, a six-month prospective chart review will be done to determine whether the clinical decision resulting from the 12-week study persisted. If a subsequent change does occur during this six-month prospective time period, the reason and rationale for the change will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* LTC residents that have been on a stable antipsychotic dose > 3 months (i.e. no changes in dose has been made during this time frame)
* Most recent RAI-MDS (Resident Assessment Instrument - Minimum Data Set) 2.0 quarterly assessment documents no change in tracked behaviours over the past 3 months while on the current on antipsychotic doses
* Power of Attorney for Healthcare (POA-HC) is locally present and able to consent
* POA-HC is proficient and can communicate fluently in English
* Chart indication for use of antipsychotic is not to manage a psychiatric condition (e.g. schizophrenia, bipolar disorder, active hallucinations and delusions)
* Currently being prescribed routine oral risperidone, olanzapine or quetiapine

Exclusion Criteria:

* Chart indication for use of antipsychotic for psychosis or other related mental health diagnoses
* POA-HC is not locally present or can not communicate fluently in English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Decision on antipsychotic dose at the end of the 12-week trial | 2 years
  Frequency and description of clinical decisions resulting from the deprescribing trial. Clinical decisions that result from this trial may include, but are not limited to, starting a lower, tapered dose, remaining on the initial starting dose, discontinuing the dose altogether, and an increased dose.

SECONDARY OUTCOMES:
Evidence for implementation in Long-Term Care | 2 years
  Rate of recruitment
Frequency of "as needed" doses used | 2 years
  The frequency of "as needed" (i.e. PRN) medications (e.g. benzodiazepines, antipsychotic, etc) used to manage behaviours. The frequency will be tracked throughout the 12 week trial and for six months after the participant has completed their trial.
Frequency of falls | 2 years
  The frequency of falls will be recorded during the 12 week trial, as well as for six months after the participant has completed the trial.
Persistence of clinical decision | 2 years
  The persistence of the clinical decision made regarding the dose of the antipsychotic by the long-term care physician and the power of attorney for personal care at six months after the participant has completed their trial.
Evidence for implementation in Long-Term Care | 2 Years
  Successful random sequence generation and allocation
Evidence for implementation in Long-Term Care | 2 Years
  Data collection from patient chart
Evidence for implementation in Long-Term Care | 2 Years
  Creation of participant summative behaviour reports
Evidence for implementation in Long-Term Care | 2 Years
  Feedback survey regarding acceptability of study rationale and procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Henry YH Siu, MSc, MD, Principal Investigator — McMaster University
Locations (1):
- Blackadar Continuing Care Centre, Dundas, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided